CLINICAL TRIAL: NCT03607643
Title: Randomized Double-Blind, Placebo-Controlled Parallel Multi-Center Study to Assess the Efficacy of Cannabidiol (BRCX014) Combined With Standard-Of-Care Treatment in Subjects With Multiple Myeloma, Glioblastoma Multiforme, and GI Malignancies
Brief Title: A Study of the Efficacy of Cannabidiol in Patients With Multiple Myeloma, Glioblastoma Multiforme, and GI Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Leaf Vertical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Olympian
Record Dates: First submitted 2018-06-05; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Cancer of Pancreas; Cancer of Liver; Cancer of Rectum; Cancer of Colon; Cancer, Gall Bladder; Myeloma Multiple; Glioblastoma Multiforme
MeSH Terms: conditions — Pancreatic Neoplasms; Liver Neoplasms; Rectal Neoplasms; Colonic Neoplasms; Gallbladder Neoplasms; Multiple Myeloma; Glioblastoma | interventions — Cannabidiol; Bortezomib; Leucovorin; Fluorouracil; Oxaliplatin; Bevacizumab; Irinotecan; Gemcitabine; Temozolomide

STUDY DESIGN:
Intervention Model Description: Study length for randomized patients in the treatment group(s) will be 180 days. For those subjects randomized into the control group(s), after 90 days of the control group study treatment, will be given the choice to rollover into the treatment group. Crossover is also permitted if there is progression of disease before 90 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, care provider, investigator, and outcomes assessor will be blinded to standard of care (SOC) alone vs treatment arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (10):
- Colon: Chemo + Placebo (Placebo Comparator): Standard of care chemotherapy for Stage IV colon or rectal cancer, will include leucovorin 350 mg/m2 IV over 2 hours Day 1, 5-FU 400 mg/m2 IV bolus followed 2400 mg/m2 IV over 46 hours, oxaliplatin 100 mg/m2 IV Day 1, bevacizumab 5 mg/kg IV day1. Irinotecan can be substituted for oxaliplatin.
  Interventions: Drug: Leucovorin; Drug: 5-FU; Drug: Oxaliplatin; Drug: Bevacizumab; Drug: Irinotecan
- Colon: Chemo + BRCX014 (Experimental): Cannabidiol (BRCX014) 200 mg daily plus Standard of care chemotherapy for Stage IV colon or rectal cancer, will include leucovorin 350 mg/m2 IV over 2 hours Day 1, 5-FU 400 mg/m2 IV bolus followed 2400 mg/m2 IV over 46 hours, oxaliplatin 100 mg/m2 IV Day 1, bevacizumab 5 mg/kg IV day1. Irinotecan can be substituted for oxaliplatin.
  Interventions: Drug: Cannabidiol; Drug: Leucovorin; Drug: 5-FU; Drug: Oxaliplatin; Drug: Bevacizumab; Drug: Irinotecan
- Rectal: Chemo + Placebo (Placebo Comparator): Standard of care chemotherapy for Stage IV colon or rectal cancer, will include leucovorin 350 mg/m2 IV over 2 hours Day 1, 5-FU 400 mg/m2 IV bolus followed 2400 mg/m2 IV over 46 hours, oxaliplatin 100 mg/m2 IV Day 1, bevacizumab 5 mg/kg IV day1. Irinotecan can be substituted for oxaliplatin.
  Interventions: Drug: Leucovorin; Drug: 5-FU; Drug: Oxaliplatin; Drug: Bevacizumab; Drug: Irinotecan
- Rectal: Chemo + BRCX014 (Experimental): Cannabidiol (BRCX014) 200 mg daily plus Standard of care chemotherapy for Stage IV colon or rectal cancer, will include leucovorin 350 mg/m2 IV over 2 hours Day 1, 5-FU 400 mg/m2 IV bolus followed 2400 mg/m2 IV over 46 hours, oxaliplatin 100 mg/m2 IV Day 1, bevacizumab 5 mg/kg IV day1. Irinotecan can be substituted for oxaliplatin.
  Interventions: Drug: Cannabidiol; Drug: Leucovorin; Drug: 5-FU; Drug: Oxaliplatin; Drug: Bevacizumab; Drug: Irinotecan
- Multiple myeloma: Chemo + Placebo (Placebo Comparator): Standard of care (SOC) chemotherapy for multiple myeloma will include a bortezomib-based regimen given at 1.3 mg/m2 on days 1, 4, 8 & 11 schedule to be repeated every 21 days.
  Interventions: Drug: Bortezomib
- Multiple myeloma: Chemo + BRCX014 (Experimental): Cannabidiol (BRCX014) 200 mg daily plus Standard of care (SOC) chemotherapy for multiple myeloma will include a bortezomib-based regimen given at 1.3 mg/m2 on days 1, 4, 8 & 11 schedule to be repeated every 21 days.
  Interventions: Drug: Cannabidiol; Drug: Bortezomib
- Pancreatic: Chemo + Placebo (Placebo Comparator): Stage IV pancreatic cancer will include a gemcitabine-based regiment at 1000 mg/m2 day 1, 7, 15 of a 21-day cycle.
  Interventions: Drug: Gemcitabine
- Pancreatic: Chemo + BRCX014 (Experimental): Cannabidiol (BRCX014) 200 mg daily plus Stage IV pancreatic cancer will include a gemcitabine-based regiment at 1000 mg/m2 day 1, 7, 15 of a 21-day cycle.
  Interventions: Drug: Cannabidiol; Drug: Gemcitabine
- GBM: Chemo + Placebo (Placebo Comparator): Standard of care chemotherapy for patients with glioblastoma multiforme includes concurrent radiation therapy (2 Gy per day for a total of 60 Gy) and temozolomide (75 mg per square meter of body-surface area per day, 7 days per week from the first to the last day of radiotherapy), followed by six cycles of adjuvant temozolomide (150 to 200 mg per square meter for 5 days during each 28-day cycle).
  Interventions: Drug: Temozolomide
- GBM: Chemo + BRCX014 (Experimental): Cannabidiol (BRCX014) 200 mg daily plus Standard of care chemotherapy for patients with glioblastoma multiforme includes concurrent radiation therapy (2 Gy per day for a total of 60 Gy) and temozolomide (75 mg per square meter of body-surface area per day, 7 days per week from the first to the last day of radiotherapy), followed by six cycles of adjuvant temozolomide (150 to 200 mg per square meter for 5 days during each 28-day cycle).
  Interventions: Drug: Cannabidiol; Drug: Temozolomide

INTERVENTIONS:
Drug: Cannabidiol — * Sublingual dose of 1 mL (0.910 g) of BRCX014 in the morning, prior to the first meal of the day
  * Sublingual dose of 1 mL (0.910 g) of BRCX014 in the afternoon, prior to the evening meal
  Other Names: BRCX014; bioRenovate CX
  Arms: Colon: Chemo + BRCX014; GBM: Chemo + BRCX014; Multiple myeloma: Chemo + BRCX014; Pancreatic: Chemo + BRCX014; Rectal: Chemo + BRCX014
Drug: Bortezomib — Standard of care (SOC) chemotherapy for multiple myeloma will include a bortezomib-based regimen given at 1.3 mg/m2 on days 1, 4, 8 & 11 schedule to be repeated every 21 days.
  Other Names: Velcade
  Arms: Multiple myeloma: Chemo + BRCX014; Multiple myeloma: Chemo + Placebo
Drug: Leucovorin — Standard of care chemotherapy for Stage IV colon or rectal cancer, will include leucovorin 350 mg/m2 IV over 2 hours Day 1, 5-FU 400 mg/m2 IV bolus followed 2400 mg/m2 IV over 46 hours, oxaliplatin 100 mg/m2 IV Day 1, bevacizumab 5 mg/kg IV day1. Irinotecan can be substituted for oxaliplatin.
  Other Names: Folinic acid
  Arms: Colon: Chemo + BRCX014; Colon: Chemo + Placebo; Rectal: Chemo + BRCX014; Rectal: Chemo + Placebo
Drug: 5-FU — Standard of care chemotherapy for Stage IV colon or rectal cancer, will include leucovorin 350 mg/m2 IV over 2 hours Day 1, 5-FU 400 mg/m2 IV bolus followed 2400 mg/m2 IV over 46 hours, oxaliplatin 100 mg/m2 IV Day 1, bevacizumab 5 mg/kg IV day1. Irinotecan can be substituted for oxaliplatin.
  Other Names: Efudex
  Arms: Colon: Chemo + BRCX014; Colon: Chemo + Placebo; Rectal: Chemo + BRCX014; Rectal: Chemo + Placebo
Drug: Oxaliplatin — Standard of care chemotherapy for Stage IV colon or rectal cancer, will include leucovorin 350 mg/m2 IV over 2 hours Day 1, 5-FU 400 mg/m2 IV bolus followed 2400 mg/m2 IV over 46 hours, oxaliplatin 100 mg/m2 IV Day 1, bevacizumab 5 mg/kg IV day1. Irinotecan can be substituted for oxaliplatin.
  Other Names: Eloxatin
  Arms: Colon: Chemo + BRCX014; Colon: Chemo + Placebo; Rectal: Chemo + BRCX014; Rectal: Chemo + Placebo
Drug: Bevacizumab — Standard of care chemotherapy for Stage IV colon or rectal cancer, will include leucovorin 350 mg/m2 IV over 2 hours Day 1, 5-FU 400 mg/m2 IV bolus followed 2400 mg/m2 IV over 46 hours, oxaliplatin 100 mg/m2 IV Day 1, bevacizumab 5 mg/kg IV day1. Irinotecan can be substituted for oxaliplatin.
  Other Names: Avastin
  Arms: Colon: Chemo + BRCX014; Colon: Chemo + Placebo; Rectal: Chemo + BRCX014; Rectal: Chemo + Placebo
Drug: Irinotecan — Standard of care chemotherapy for Stage IV colon or rectal cancer, will include leucovorin 350 mg/m2 IV over 2 hours Day 1, 5-FU 400 mg/m2 IV bolus followed 2400 mg/m2 IV over 46 hours, oxaliplatin 100 mg/m2 IV Day 1, bevacizumab 5 mg/kg IV day1. Irinotecan can be substituted for oxaliplatin.
  Other Names: Camptosar
  Arms: Colon: Chemo + BRCX014; Colon: Chemo + Placebo; Rectal: Chemo + BRCX014; Rectal: Chemo + Placebo
Drug: Gemcitabine — Stage IV pancreatic cancer will include a gemcitabine-based regiment at 1000 mg/m2 day 1, 7, 15 of a 21-day cycle.
  Other Names: Gemzar
  Arms: Pancreatic: Chemo + BRCX014; Pancreatic: Chemo + Placebo
Drug: Temozolomide — Standard of care chemotherapy for patients with glioblastoma multiforme includes concurrent radiation therapy (2 Gy per day for a total of 60 Gy) and temozolomide (75 mg per square meter of body-surface area per day, 7 days per week from the first to the last day of radiotherapy), followed by six cycles of adjuvant temozolomide (150 to 200 mg per square meter for 5 days during each 28-day cycle).
  Other Names: Temodar
  Arms: GBM: Chemo + BRCX014; GBM: Chemo + Placebo

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Parallel, Multi-Center Study to Assess the Efficacy of BRCX014 Combined with Standard-Of-Care Treatment in Subjects with Glioblastoma Multiforme, Multiple Myeloma, and GI Malignancies

DETAILED DESCRIPTION:
Several studies have shown a potential anti-tumor role for cannabinoids by modulating cell signaling pathways, inhibiting angiogenesis, inducing apoptosis, and overcoming chemotherapy resistance. In phase I trials, cannabinoids have been shown to enhance the uptake of chemotherapy into malignant cells without affecting normal cells. The investigators seeks to demonstrate that the combination of chemotherapy with BRCX014 will have a greater anti-tumor and anti-proliferative activity when compared to standard of care alone.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent
2. Male and Females age 18 to 80 years old at the time of screening
3. Confirmed tissue diagnosis of Multiple myeloma, GI malignancy by a licensed pathologist
4. A performance status 0-1 on the Eastern Cooperative Oncology Group (ECOG) scale.
5. Females of childbearing potential willing to utilize two approved forms of contraceptives (e.g., birth control, abstinence, spermicidal lube, intrauterine device [IUD])
6. Male study subjects must be willing to use two approved forms of contraceptives (e.g., physical barrier-condoms, abstinence, spermicidal lube)

Exclusion Criteria:

1. Subject is pregnant or plans to become pregnant or actively lactating/nursing
2. Hypersensitivity to any ingredient in the study product
3. Initial laboratory values as determined by the principal investigator to be clinically significant
4. A substance abuse history within the last five years
5. Any diseases or conditions that may interfere with the conduct of the study or interpretation of the study results
6. .Close affiliation with the investigational site (e.g., a close relative of the investigator), dependent person (employee or student of investigational site, or sponsor's staff)
7. Currently enrolled in another investigational clinical study
8. A known history of severe depression or psychiatric disorders or active suicidal ideation
9. Inability or unwillingness to cooperate with the study procedures for any reasons

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-01-15 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Response rate | Through study completion, an average of one year
  The primary objective of this study is to evaluate the overall response rates of cancer patients as assessed by standard criteria.

SECONDARY OUTCOMES:
Time to progression (TTP) in patients using lab results and radiographic data. | Through study completion, an average of one year
  A secondary objective of this study is to measure TTP using lab results and radiographic data.
Progression-free survival (PFS) in patients using lab results and radiographic data. | Through study completion, an average of one year
  A secondary objective of this study is to measure PFS using lab results and radiographic data.
Quality-of-life assessment in patients using patient-reported outcomes (PRO) data. | Through study completion, an average of one year
  A secondary objective of this study is to collect patient-reported outcomes (PRO) data.
Quality-of-life assessment in patients using clinician-reported outcomes (ClinRO) data. | Through study completion, an average of one year
  A secondary objective of this study is to collect clinician-reported outcomes (ClinRO) data.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah F Katta, DO, Principal Investigator — Leaf Vertical Inc.
Locations (1):
- Southwest Cancer Center, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No